CLINICAL TRIAL: NCT04300374
Title: Effects of Remifentanil Infusion on Emergence Delirium After Dental Surgery in Children
Status: Completed | Type: Observational
Sponsor: Erzincan University (Other)
Responsible Party: Principal Investigator, Nurcan Kutluer Karaca, Assistant Professor, Erzincan University
Other Study IDs: Erzincan Universty
Record Dates: First submitted 2019-11-08; First posted 2020-03-09 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Emergence Delirium
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Sevoflurane only: inhalation of sevoflurane during general anesthesia
  Interventions: Other: The Paediatric Anaesthesia Emergence Delirium scale assesment which was recorded postoperatively
- Remifentanil and Sevoflurane: remifentanil infusion and inhalation of sevoflurane during general anesthesia
  Interventions: Other: The Paediatric Anaesthesia Emergence Delirium scale assesment which was recorded postoperatively

INTERVENTIONS:
Other: The Paediatric Anaesthesia Emergence Delirium scale assesment which was recorded postoperatively — routine remifentanil infusion during general anesthesia

SUMMARY:
In this study, the investigators tried to show the effect of remifentanil on emergence delirium caused by sevoflurane used in general anesthesia.We planned a retrospective study. We formed two groups of 80 participants. One group included patients who were received remifentanil infusion during general anesthesia.The other group included patients who were received only sevoflurane inhalation anesthesia.

The patients included in the study were evaluated for emergence delirium in the postoperative period be evaluating the past recorded informations.

ELIGIBILITY:
Inclusion Criteria American Society of Anesthesiologists score 1-2

-

Exclusion Criteria:

* neurological disease, psychiatric illness

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: All patients between 2 and 6 years old having American Society of Anesthesiologists score 1-2.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
emergence delirium | 30 minute after operation
  incidence of emergence delirium

CONTACTS AND LOCATIONS:
Locations (1):
- Nurcan Kutluer Karaca, Erzincan, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No